CLINICAL TRIAL: NCT01100788
Title: Satiety Response of Short Chain Fructooligosaccharide
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Joanne Slavin, University of Minnesota
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 0806M37444
Record Dates: First submitted 2010-03-05; First posted 2010-04-09 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
MeSH Terms: interventions — fructo-oligosaccharide-shitake

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): No treatment
  Interventions: Other: Placebo
- scFOS 5 g (Experimental): 5 g scFOS
  Interventions: Dietary Supplement: Short chain fructo-oligosaccharide (scFOS) 5 g
- scFOS 8 g (Experimental): 8 g scFOS
  Interventions: Dietary Supplement: Short chain fructooligosaccharide (scFOS) 8 g

INTERVENTIONS:
Dietary Supplement: Short chain fructo-oligosaccharide (scFOS) 5 g — Dietary Supplement: scFOS 5 g
  Novel fiber administered in two 5 g doses--the first in a beverage and the second in a solid chew.
  Other Names: fructo-oligosaccharide
  Arms: scFOS 5 g
Other: Placebo — Treatment without scFOS fiber
  Arms: Placebo
Dietary Supplement: Short chain fructooligosaccharide (scFOS) 8 g — Novel fiber administered in two 8 g doses--the first in a beverage and the second in a solid chew.
  Arms: scFOS 8 g

SUMMARY:
Populations that report high fiber consumption demonstrate lower rates of obesity. Enhanced satiety may play a key role in this relationship. The colonic fermentation of fibers is theorized to influence satiety and food intake. Short chain fructooligosaccharide (scFOS) are rapidly fermentable fibers that can easily be added to foods to impact these parameters.

The objective of this study was to evaluate the satiety response of scFOS and its ability to decrease food intake.

DETAILED DESCRIPTION:
Intervention study with fiber added to beverages and acute effects on satiety measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18-64 years
* Non-smoking
* Not taking medication
* Non-dieting (weight stable in prior 3 months)
* BMI 18-27
* English literacy

Exclusion Criteria:

* Do not regularly consume breakfast
* Food allergies to ingredients found in study products
* BMI <18 or >27
* Diagnosed cardiovascular, renal, or hepatic disease diabetes mellitus
* Cancer in previous 5 years (except basal cell carcinoma of the skin)
* Any gastrointestinal disease or condition
* Recent bacterial infection (< 3 months)
* Recent or concurrent participation in an intervention research study
* History of drug or alcohol abuse in prior 6 months
* Use of lipid-lowering, anti-hypertensive, or anti-inflammatory steroid medication
* Eating disorder
* Vegetarians
* People who eat more than approximately 15 grams of fiber per day
* Women who are pregnant or lactating
* Women with irregular menstrual cycles

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Satiety response using visual analogue scales | 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).

SECONDARY OUTCOMES:
Ad libitum food intake | 240 minutes postprandially and over 24 hours
Breath hydrogen response | 0, 240 minutes
Gastrointestinal tolerance using visual analogue scales (VAS) | 24 hours
  Subjective ratings of bloating, stool consistency, and flatulence on VAS. A stool count was also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States